CLINICAL TRIAL: NCT06381323
Title: Study on the Clinical Efficacy and Safety of the New Mineralocorticoid Receptor Antagonist Finerenone in the Treatment of Primary Aldosteronism: a Multicenter, Prospective, Open-label Clinical Study
Brief Title: The Clinical Efficacy and Safety of Finerenone in the Treatment of Primary Aldosteronism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA2024
Record Dates: First submitted 2024-04-16; First posted 2024-04-24 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-03

CONDITIONS: Primary Aldosteronism; Finerenone; Mineralocorticoid Receptor Antagonist
Keywords: Primary Aldosteronism; Finerenone; Mineralocorticoid Receptor Antagonist; Hypertension; 24-hour ambulatory blood pressure monitoring; Daytime SBP
MeSH Terms: conditions — Hyperaldosteronism; Hypertension | interventions — finerenone; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Finerenone (Experimental): Recruitment of diagnosed patients with PA from multiple centers, confirmation of subject eligibility according to inclusion criteria and exclusion criteria, and signing of informed consent forms. All eligible subjects enter a 2-week enrollment phase and only take stable doses of controlled-release nifedipine. After completing baseline examinations, subjects with SBP <180 and ≥140 mmHg and DBP <120 and ≥90 mmHg enter the follow-up phase of the treatment period. Eligible subjects receive a starting dose of 20 mg qd of Finerenone. If the blood pressure is still ≥140/90 mmHg at week 4, serum potassium is <5.0 mmol/L, and eGFR has decreased <30% compared to baseline, the Finerenone dose is adjusted to 40 mg qd.
  Interventions: Drug: Finerenone

INTERVENTIONS:
Drug: Finerenone — All eligible subjects enter a 2-week enrollment phase and only take stable doses of controlled-release nifedipine. After completing baseline examinations, subjects with SBP <180 and ≥140 mmHg and DBP <120 and ≥90 mmHg enter the follow-up phase of the treatment period. Eligible subjects receive a starting dose of 20 mg qd of Finerenone. If the blood pressure is still ≥140/90 mmHg at week 4, serum potassium is <5.0 mmol/L, and eGFR has decreased <30% compared to baseline, the Finerenone dose is adjusted to 40 mg qd.
  Other Names: Nifedipine

SUMMARY:
The purpose of our research is to clarify the therapeutic efficacy and safety of Finerenone in patients with Primary Aldosteronism and explore the effective clinical predictive indicators of Finerenone in the treatment of Primary Aldosteronism.

DETAILED DESCRIPTION:
Primary aldosteronism(PA) is a clinical syndrome characterized by autonomous aldosterone secretion in the body caused by adrenal cortical adenoma or hyperplasia not regulated by renin, angiotensin II, and sodium status regulation. It is the most common cause of secondary hypertension, accounting for about 10% of all hypertensive patients. The latest prospective study in China showed that the prevalence of primary aldosteronism in newly diagnosed hypertensive patients was 4%, with an additional 3% of suspicious primary aldosteronism patients. Excessive activation of the mineralocorticoid receptor (MR) in the body leads to well-known increased circulating volume overload, hypertension, and hypokalemia, as well as significantly increased cardiovascular, renal, and mortality risks. Therefore, primary aldosteronism is currently considered a new public health problem and has important implications for early diagnosis and precise treatment of primary aldosteronism.

Only about 30% of patients with PA (aldosterone-producing adenoma or unilateral adrenal hyperplasia) can be cured or relieved through surgical resection, while about 65% of patients with primary aldosteronism caused by bilateral adrenal cortical hyperplasia require drug treatment. Currently, the only available drug in China is the first-generation mineralocorticoid receptor antagonist, spironolactone, which is greatly limited in its use due to its significant side effects on the gonads caused by the blockade of androgens and progesterones. Another MRA, eplerenone, which has not yet been marketed in China, is expensive and clinically inferior to spironolactone. Therefore, a large number of patients with primary aldosteronism are currently not using or using low doses of spironolactone, unable to fully counteract the high aldosterone effect, and unable to effectively control the risk of cardiovascular and renal damage. Therefore, it is necessary to explore new drugs for the treatment of primary aldosteronism.

Finerenone is a newly developed novel non-steroidal MRA, which has higher affinity and selectivity for MR binding compared to steroidal MRA (spironolactone or eplerenone). Existing clinical research results suggest that Finerenone can effectively reduce the risk of cardiovascular and renal damage in patients with chronic kidney disease and diabetes, and has good safety.

This study aims to be the first internationally to conduct clinical research on the use of the novel mineralocorticoid receptor antagonist finerenone for the treatment of primary aldosteronism. Through a multicenter, prospective, open-label study, the clinical efficacy and safety of this medication will be clearly established, providing high-level evidence of the use of finerenone in patients with primary aldosteronism. The project's results will offer a new option for the pharmacological treatment of primary aldosteronism, with the goal of better controlling patients' biochemical abnormalities, effectively reducing the risk of cardiovascular and renal damage, and improving disease prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-75 years old.
2. History of hypertension, with a sitting SBP ≥140 and <180 mmHg, and a sitting DBP ≥90 and <120 mmHg during the last two evaluations within the observation period.
3. Patients with PA who are eligible for drug treatment.
4. Diagnostic criteria for primary aldosteronism: (1) Hypertension or use of antihypertensive medications, with or without hypokalemia; (2) Screening test: Baseline plasma aldosterone to renin ratio (ARR) >30 (ng/dl)/(ng/ml/h) or ARR >2.4 (ng/dl)/(mU/L), with plasma aldosterone >15 ng/dl and plasma renin activity <1.0 ng/ml/h; (3) At least one confirmed test is positive: ① After a captopril test, plasma aldosterone decreases by <30% or plasma aldosterone is ≥11 ng/dl, with suppressed renin activity; ② Sitting saline infusion test results in a plasma aldosterone ≥10 ng/dl.
5. eGFR ≥60 ml/ (min*1.73m2).
6. Signed informed consent form.

Exclusion Criteria:

1. Other secondary hypertension (such as renal vascular hypertension, Cushing's syndrome, subclinical Cushing's syndrome, and pheochromocytoma) or hypertensive crisis.
2. Orthostatic hypotension.
3. Heart failure, acute myocardial infarction, stroke, transient ischemic attack, or other acute cardiovascular events within the past 6 months.
4. History of adrenal surgery within the past 6 months.
5. History of carotid artery surgery within the past 6 months.
6. History of arterial vascular reconstruction surgery within the past 6 months.
7. Hospitalization within the past year due to severe hyperkalemia, with serum potassium levels <2.5 or ≥5.0 mmol/L.
8. Abnormal liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5× upper limit of normal (ULN), total bilirubin (TBIL) > 1.5× ULN.
9. Use of spironolactone, hydralazine, or minoxidil within 30 days prior to enrollment.
10. Concurrent use of potent CYP3A4 inhibitors or inducers for treatment.
11. Known or suspected tumors; other autoimmune diseases, uncontrolled infectious diseases, severe respiratory, blood, and neurological diseases.
12. Pregnancy or planning pregnancy within 3 months before or after treatment, and breastfeeding women.
13. Mental illness, alcohol or drug abuse, inability to cooperate with treatment.
14. Patients with pacemakers.
15. Participation in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
24h systolic BP drop value | 12 weeks
  The average daytime systolic blood pressure drop from baseline levels after treatment with Finerenone at 12 weeks.

SECONDARY OUTCOMES:
The change of diastolic BP from the baseline level after Finerenone treatment | Baseline,4 weeks,8 weeks,12 weeks,16 weeks
  To Clarify the antihypertensive effect of Finerenone by measuring daytime diastolic blood pressure from baseline to the end of treatment .
Hypertension remission rate | Baseline,4 weeks,8 weeks,12 weeks,16 weeks
  The proportion of patients with SBP<140mmHg and DBP<90mmHg.
Change of serum potassium level | Baseline,4 weeks,8 weeks,12 weeks,16 weeks
  Proportion of patients with normal blood potassium levels (serum potassium level ≥ 3.5mmol/L and ≤ 5.5mmol/L).
Change of plasma renin activity | Baseline,4 week,8 weeks,12 weeks,16 weeks
  to compare plasma renin activity during the progression
Change of ARR | Baseline,4 weeks,8 weeks,12 weeks,16 weeks
  To see if Finerenone can influence ARR[(ng/dl)/(ng/ml/h)]
Change of UACR | Baseline,4 weeks,8 weeks,12 weeks,16 weeks
  Compared to the placebo group, the risk of kidney disease progression in patients with type 2 diabetes and chronic kidney disease decreased by 18% after treatment with nonnarcotic ketones.
Change of eGFR | Baseline,4 weeks,8 weeks,12 weeks,16 weeks
  Estimated glomerular filtration rate (eGFR) decline condition.

OTHER OUTCOMES:
Incidence of Treatment-Adverse Events as assessed by gynaecomastia, mastodynia, menstrual abnormalities, impotence, hyperkalemia and other adverse events. | Baseline,4 weeks,8 weeks,12 weeks,16 weeks
  1. Adverse effects such as gynaecomastia, mastodynia, menstrual abnormalities and impotence due to its agonist activity.
  2. Hyperkalemia.
  3. Other adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Li, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Department of Endocrinology, Drum Tower Hospital affiliated to Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.

REFERENCES:
- [Derived] Li P, Yang F, Lou Y, Zhang Z, Du Y, Zhang J, Ren Y, Tong A, Xie Z, Shi B, Liu J, Liu L, Zhu D. Efficacy and Safety of Finerenone in Patients With Primary Aldosteronism: A Multicenter Prospective Study. Hypertension. 2026 Jan 22. doi: 10.1161/HYPERTENSIONAHA.125.26048. Online ahead of print. PMID 41568520